CLINICAL TRIAL: NCT02486120
Title: Are Genetic Counselors Screening Adolescents for Suicide Risk? A Mixed Methods Study
Brief Title: Are Genetic Counselors Screening for Adolescent Suicide Risk?
Status: Completed | Type: Observational
Sponsor: National Human Genome Research Institute (NHGRI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999915152; 15-HG-N152
Record Dates: First submitted 2015-06-30; First posted 2015-07-01 (Estimated); Last update posted 2019-10-23 (Actual); Status verified 2017-05-24

CONDITIONS: Healthy Volunteers
Keywords: Genetic Counseling; Clinical Decision-Making

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional

SUMMARY:
Background:

- Suicide is one of the main causes of death for adolescents in the U.S. The most effective way to decrease suicide is by training doctors to recognize the risk factors in their clients. One risk factor for suicide is chronic illness. So pediatric genetic counselors come across high-risk clients. But the suicide risk assessment (SRA) practices of these counselors are not well known. Researchers want to study learn more about this.

Objectives:

- To describe the practices, attitudes, and beliefs of genetic counselors about SRA of adolescents.

Eligibility:

- Genetic counselors who see adolescents ages 10 21

Design:

* A study will be open to a listserv for genetic counselors.
* Participants will take a survey on their own.
* The survey will be online on a secure website.
* Participants will give data about themselves. This can include age, gender, job, etc.
* The survey will be about 60 questions.
* The survey will take around 20 25 minutes.
* The questions are about participants experiences, practices, attitudes, and beliefs about SRA.

DETAILED DESCRIPTION:
This study proposes to describe the practices, attitudes, and beliefs of genetic counselors in relation to suicide risk assessment (SRA) of their adolescent clients. Suicide is a major public health issue and one of the leading causes of death for adolescents in the U.S. Analysis of suicide prevention campaigns has shown that the most effective way to decrease suicide is by training physicians to recognize suicide risk factors in their patients . However, pediatricians do not consistently screen youth for suicide risk during routine check-ups. As chronic illness is an additional risk factor for suicide, pediatric genetic counselors encounter particularly high-risk clients and are well-positioned to assess for suicide risk due to the psychosocial nature of their work. However, the SRA practices of genetic counselors are largely unknown. In this study, the Transtheoretical Model of Behavior Change is used as a framework to describe how genetic counselors SRA self-efficacy and perceptions of the pros and cons of SRA relate to stages of readiness and practices of assessing clients for suicide risk. Specifically, we will be surveying genetic counselors about their practices, attitudes and beliefs concerning SRA of adolescent clients. First, we will determine genetic counselors frequency of SRA and their stage of readiness for routine screening. Second, we will measure genetic counselors SRA self-efficacy and their perceptions of the pros and cons of screening their clients. We will examine whether self-efficacy and perceptions of pros and cons are predictors of genetic counselors stage of readiness for routine suicide screening. Finally, we will qualitatively assess genetic counselors perceptions of the usability of a validated suicide screening tool (the ASQ) in genetic counseling sessions and their interest in receiving suicide screening training. We will use a cross-sectional, mixed-methods design in which counselors will complete an online questionnaire with quantitative components and open-ended responses. Participants will be recruited through the National Society of Genetic Counselors Student Research Survey listserv.

ELIGIBILITY:
* INCLUSION CRITERIA:

Participants in this study will be English speaking women and men who are graduates of accredited genetic counseling programs. Those who currently or within the past year have worked in-person with adolescent patients between the ages of 10 and 21 may be included in the survey.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 267 (Actual)
Dates: Start 2015-06-22; Primary Completion 2016-05-31 (Actual); Study Completion 2017-05-24 (Actual)

PRIMARY OUTCOMES:
Previous performance of adolescent patient suicide risk assessment | Ongoing

CONTACTS AND LOCATIONS:
Overall Officials: Lori Erby, Ph.D., Principal Investigator — National Human Genome Research Institute (NHGRI)
Locations (1):
- National Human Genome Research Institute (NHGRI), 9000 Rockville Pike, Bethesda, Maryland, United States